CLINICAL TRIAL: NCT06155136
Title: Real-world Evidence on Patients With Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC) Long-term Survival After Treatment With Liposomal Irinotecan (NALLONG)
Brief Title: RWE on Patients With mPDAC Long-term Survival After Treatment With Liposomal Irinotecan
Acronym: NALLONG
Status: Active, not recruiting | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-95013-001-INT
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to describe mPDAC patients still alive one year after the first cycle of nal-IRI

DETAILED DESCRIPTION:
The objectives on patients still alive one year after the first cycle of nal-IRI :

* Characterize mPDAC patient population according to their demographics
* Identify PDAC treatment by line of treatment from diagnosis to last treatment
* Explore prognostic factors of longer Overall Survival (OS) and Progression Free Survivor (PFS) among mPDAC patients showing long-term Survival

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years (≥ 19 years in South Korea)
* Cytologically confirmed mPDAC at initiation of the nal-IRI treatment
* All patients receiving a nal-IRI + 5-flurouracil/leucovorin regimen should have been pre-treated with a gemcitabine-based regimen
* Initiation of a systemic therapy with nal-IRI (index date) during the study eligibility period (between January 1, 2018, and December 31, 2021)
* At least one cycle of nal-IRI-containing regimen should have been administered
* A minimum 1-year survival from the index date (initiation date of nal-IRI-containing regimen)
* Availability of data related to survival outcomes in the patient medical record
* Patients deceased or not at the time of enrollment will be eligible for inclusion in the study

Exclusion Criteria:

* No documentation of systemic therapy outcomes or prior treatments in patient medical records
* Patients with second concomitant metastatic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients still alive one year after the initiation of NAliri
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Disease characteristic according to age | Through study completion (approximatively 5 months)
  Tumor stage (localized/locally advanced/metastatic)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum der Universität München, - Anstalt des öffentlichen Rechts -, Munich, Germany